"CLINICAL-INSTRUMENTAL EVALUATION OF THE EFFICACY OF A DIETARY SUPPLEMENT CLAIMING ANTIHAIR LOSS PROPERTIES Double-blind, randomized, placebo-controlled, multicentric study".

**Protocol ID:** IT0006736/24

**Date:** 06Dec2024

## Study synopsis

The study is aimed to assess the efficacy of a dietary supplement in two different formulations (capsules and drinkable supplements) claimed to reduce hair loss in female and male subjects showing androgenetic alopecia (AGA) or chronic telogen effluvium.

In order to reach this goal a randomized, double-blind, parallel groups, placebo-controlled study was carried out on 240 (264 enrolled) healthy female and male subjects included according to specific inclusion and non-inclusion criteria. In particular, male and female subjects aged between 18 and 62 years old, including at least 70% of female subjects aged over 30 years old. 50% of the subjects showed chronic telogen effluvium and 50% of subjects showed androgenetic alopecia (AGA). As per randomization list the subjects were assigned to one of the following study groups: dietary supplement capsule, dietary supplement capsule placebo, dietary supplement drinkable and dietary supplement drinkable placebo. The subjects used assigned product once a day during 6 months with safety and efficacy evaluations at baseline, 3 months (3M) and 6 months (6M) of product use. The study was approved by an independent ethics committee.